CLINICAL TRIAL: NCT02304107
Title: Comparison Between Letrozole and Urinary Purified FSH in Women With Clomiphene Citrate Resistant Polycystic Ovarian Syndrome: A Randomised Controlled Trial
Brief Title: Comparison Between Letrozole and Urinary Purified FSH in Women With Clomiphene Citrate Resistant Polycystic Ovarian Syndrome.
Acronym: FSH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sub 6
Record Dates: First submitted 2014-11-26; First posted 2014-12-01 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FSH (Active Comparator): 70 women will receive urinary purified FSH (Fostimon® IBSA, Switzerland) 75IU daily for 7 days starting from the 3rd day of menstruation or progesterone withdrawal bleeding. If the follicle does not exceed 9 mm the dose will be increased by 37.5 IU every 7 days.
  Interventions: Drug: FSH
- Letrozole (Active Comparator): 70 women will receive Letrozole (Femara®, Novartis, Switzerland) 2.5mg twice daily for 5 days starting from the 3rd day of menstruation or progesterone withdrawal bleeding.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: FSH — 75IU daily for 7 days starting from the 3rd day of menstruation or progesterone withdrawal bleeding. If the follicle does not exceed 9mm the dose will be increased by 37.5IU every 7 days
  Arms: FSH
Drug: Letrozole — 70 women will receive Letrozole (Femara®, Novartis, Switzerland) 2.5mg twice daily for 5 days starting from the 3rd day of menstruation or progesterone withdrawal bleeding.
  Arms: Letrozole

SUMMARY:
210 women with clomiphene resistant PCOS will be randomly divided into 3 equal groups using computer generated random numbers. Group 1 will receive FSH, group 2 will have Letrozole and group 3 will act as the control group with no intervention.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in reproductive age, with an incidence of 5 -10%. Classically clomiphene citrate (CC) is the first approach to induce ovulation in patients with PCOS. Although 70-80% of PCOS women can ovulate by the treatment with CC, only 40%of the PCOS women become pregnant. Women who do not ovulate with increasing doses of CC are described as being CC-resistant and remain a major challenge in gynecologic endocrinology. Traditional alternatives for CC-resistant patients include gonadotropin therapy and laparoscopic ovarian diathermy.

Gonadotropin therapy is widely used for ovulation induction in CC-resistant PCOS patients. The use of purified FSH preparation virtually free of LH activity, is a recommendable treatment since there is evidence that pure FSH may significantly reduce tonic LH levels, favourably alter the intraovarian hormonal milieu, and promote the initial follicular development with minimal risk of multiple follicular growth or ovarian hyperstimulation.

The use of metformin in PCOS is associated with cycle regulation, improved ovulation, and a reduction in circulating androgen levels. Metformin likely plays its role in improving ovulation induction in women with PCOS through a variety of actions, including reducing insulin levels and altering the effect of insulin on ovarian androgen biosynthesis, theca cell proliferation, and endometrial growth. In addition, potentially through a direct effect, it inhibits ovarian gluconeogenesis and thus reduces ovarian androgen production.

Letrozole is an orally-active aromatase inhibitor, with good potential for ovulation induction. Letrozole acts by reducing estrogen production by blocking androgens to estrogens conversion. Additionally, it has no adverse effect on endometrium and cervical mucus (7). This releases the pituitary from negative feedback of estrogens and releases FSH. Also, an added positive effect is increased follicular sensitivity to FSH through amplification of FSH receptor gene expression.

Hyper-insulinemia, which is closely associated with PCOS, is thought to be one of the causative factors for CC resistance. The prevalence of insulin resistance in PCOS is close to 50%.

All women with clomiphene resistant PCOS attending the subfertility clinic of Cairo university hospitals will be invited to participate in the study. PCOS diagnosis will be based on chronic anovulation and sonographic picture of polycystic ovaries (10). Clomiphene resistance will be defined as failure of ovulation in spite of receiving 150mg of clomiphene citrate for 5 days during the menstrual cycle.

Exclusion criteria are age >40 years, other causes of infertility, hperprolactinaemia, allergy to FSH or metformin, previous FSH or LOD therapy, and body mass index (BMI)>35.

The study will be explained to all the participants and a written informed consent will be obtained before participation.

Full history will be taken followed by complete examination and sonographic evaluation. Sonographic picture of polycystic ovaries will be defined when there are at least 12 follicles 2-9mm in the ovary and/or ovarian volume>10cm3 (10) 210 women with clomiphene resistant PCOS will be randomly divided into 3 equal groups using computer generated random numbers. Group 1 will receive FSH, group 2 will have Letrozole and group 3 will act as the control group with no intervention.

Group 1 will receive urinary purified FSH (Fostimon® IBSA, Switzerland) 75IU daily for 7 days starting from the 3rd day of menstruation or progesterone withdrawal bleeding. If the follicle does not exceed 9mm the dose will be increased by 37.5IU every 7 days. The cycle will be cancelled if no follicles exceed 9mm 4 weeks after starting FSH. Group 2 will receive Letrozole (Femara®, Novartis, Switzerland) 2.5mg twice daily for 5 days starting from the 3rd day of menstruation or progesterone withdrawal bleeding.

Group 3 will have regular progesterone withdrawal bleeding in the form of norethisterone (stereonate® Hi Pharm, Egypt).

Serial vaginal ultrasound scans were done starting from the 10th day of menstruation, the frequency of monitoring will be individualized according to the women's response. When the dominant follicle reaches 17mm or more women will receive Human chorionic gonadotrophin (Choriomon® IBSA, Switzerland) 5000IU and a timed intercourse will be advised 36 hours later.

ELIGIBILITY:
Inclusion Criteria:

* Clomiphene resistant PCOS.

Exclusion Criteria:

* Other causes of infertility.
* Hyperprolactinaemia.
* Allergy to Letrozole or FSH.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2013-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Ovulation | 6 weeks after starting the intervention
  Regular vaginal ultrasounds will be done starting from the 8th day of starting the drug.

SECONDARY OUTCOMES:
Pregnancy | 6 months after starting the intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - BeniSuef University hospitals, BeniSuef
  - Cairo University Hospitals, Cairo

REFERENCES:
- [Background] Kar S. Clomiphene citrate or letrozole as first-line ovulation induction drug in infertile PCOS women: A prospective randomized trial. J Hum Reprod Sci. 2012 Sep;5(3):262-5. doi: 10.4103/0974-1208.106338. PMID 23531705
- [Background] Vendola K, Zhou J, Wang J, Famuyiwa OA, Bievre M, Bondy CA. Androgens promote oocyte insulin-like growth factor I expression and initiation of follicle development in the primate ovary. Biol Reprod. 1999 Aug;61(2):353-7. doi: 10.1095/biolreprod61.2.353. PMID 10411511
- [Derived] Hassan A, Shehata N, Wahba A. Cost effectiveness of letrozole and purified urinary FSH in treating women with clomiphene citrate-resistant polycystic ovarian syndrome: a randomized controlled trial. Hum Fertil (Camb). 2017 Apr;20(1):37-42. doi: 10.1080/14647273.2016.1242783. Epub 2016 Nov 8. PMID 27825272